CLINICAL TRIAL: NCT06054841
Title: Reshaping Postpartum Follow-up in Women With High Risk Pregnancies
Brief Title: Reshaping Postpartum Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006037
Record Dates: First submitted 2023-05-22; First posted 2023-09-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hypertension in Pregnancy; Gestational Diabetes; Cervical Dysplasia
Keywords: Postpartum followup; hypertensive disorders of pregnancy; eclampsia; pre-eclampsia; pap smear; gestational diabetes
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Diabetes, Gestational; Uterine Cervical Dysplasia; Eclampsia; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow up cards (Experimental): Subjects will receive a personalized postpartum health card with recommendations for follow up based on their comorbid conditions in pregnancy. They will receive education about these comorbid conditions when they receive their cards.
  Interventions: Behavioral: Postpartum follow up card
- Standard education (Placebo Comparator): Subjects will receive standard postpartum education as it is routinely performed by nurses prior to discharge.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Postpartum follow up card — The intervention will consist of a card given to patients at time of discharge. One side of the card will list the patient's name and a list of recommended postpartum follow-up appointments based on their diagnoses at the time of discharge. The back of the card will list relevant phone numbers to assist patients with scheduling.
  Arms: Follow up cards
Other: Control — No deviation from standard discharge education
  Arms: Standard education

SUMMARY:
The aim of this study is to evaluate the impact of personalized postpartum follow-up cards on completion of postpartum health related tasks. The intervention will consist of a card given to patients at time of discharge. One side of the card will list the patient's name and a list of recommended postpartum follow-up appointments based on their diagnoses at the time of discharge. Participants will be randomized to this intervention or the control group, which will consist of standard education routinely given at discharge.

The primary endpoint will be the rate of completion of a postpartum blood pressure check or two hour glucose tolerance test, or both, depending on the patient's discharge diagnosis within the first year after discharge. The secondary endpoints will include establishing care with a primary care provider within the first year after delivery, or completion of postpartum pap smear or colposcopy, as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >=18 years of age
* Ability to read English or Spanish
* Delivered via vaginal delivery or c-section within the past 48 hours
* Able to consent for themselves

Exclusion Criteria:

* Received antepartum care at a facility outside of the Medstar system or plans to continue care with a facility outside of the Medstar system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure check | 6 months
  Rate of attendance at a blood pressure check one week postpartum
Two hour glucose tolerance test | 6 months
  Rate of completion of two hour glucose tolerance test at six weeks postpartum

SECONDARY OUTCOMES:
Cervical cancer screening | 6 months
  Rate of completion of postpartum pap smear or colposcopy as indication
Primary care | 6 months
  Rate of attendance at visit with primary care provider for annual exam

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No